CLINICAL TRIAL: NCT05722951
Title: Metformin Efficacy and Safety in Epileptic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Omnia Ashraf Abd El Aziz Ahmed, Teacher Assisstant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107353
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam; Valproic Acid; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (+ve control) (Active Comparator): levetiracetam &/or sodium valproate
  Interventions: Drug: Levetiracetam &/or sodium valproate
- Treatment group (Experimental): metformin + (levetiracetam &/or sodium valproate)
  Interventions: Drug: Levetiracetam &/or sodium valproate; Drug: Metformin

INTERVENTIONS:
Drug: Levetiracetam &/or sodium valproate — levetiracetam &/or sodium valproate will be given to 30 patients and monitored for 6 months
  Other Names: Levetiracetam &/or valproic acid
Drug: Metformin — metformin + (levetiracetam &/or sodium valproate) will be given to 30 patients and monitored for 6 months will be given to 30 patients and monitored for 6 months
  Arms: Treatment group

SUMMARY:
The goal of this clinical trial is to Evaluating Metformin Efficacy and Safety when Co-administered with Antiepileptic Drugs in Patients with Seizures. The main question it aims to answer is:

* Does metformin have beneficial effect on epileptic patients?
* How metformin can affect epileptic patient's health?

Participants will be divided into 2 groups (control group and treatment group)

* Control group will receive standard treatment (levetiracetam &/or sodium valproate).
* Treatment group will receive standard treatment (levetiracetam &/or sodium valproate) + metformin

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old
* Obese and overweight patients with body mass index (BMI) ≥ 25.
* Diabetic & non diabetic patients.

Exclusion Criteria:

* Patients with severe liver damage or kidney disease (eGFR below 45mL/min/1.73 m²).
* Patients having acute or chronic disease which may cause tissue hypoxia and increase the risk of lactic acidosis (e.g. cardiac/respiratory failure, recent myocardial infarction).
* Patients who are already taking metformin.
* Cancer patients.
* Pregnant or lactating women.
* Patients with known hypersensitivity to the drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Seizures Frequency | 6 months
  will be recorded using seizures diary.
Seizures Severity | 6 months
  will be measured using chalfont seizures severity scale.
Quality of Life level | 6 months
  will be recorded using SF-36 health survey.

SECONDARY OUTCOMES:
Change in BMI | 6 months
Change in biological markers | 6 months
  eg. serum lactate.

CONTACTS AND LOCATIONS:
Locations (1):
- Omnia Ashraf Abd El Aziz Ahmed Kotb, Alexandria, Egypt